CLINICAL TRIAL: NCT04826471
Title: Multicenter, Open Label, Uncontrolled Clinical Investigation on the Performance and Safety of DermoRelizema Ecofoam in the Management of Some Dermatitis in the Adult
Brief Title: Clinical Investigation on the Performance and Safety of DermoRelizema Ecofoam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Relife S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ReGl/20/Dec-Der/001
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Results first posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-01

CONDITIONS: Dermatitis
Keywords: ecofoam; DermoRelizema ecofoam; dermatitis treatment; mild moderate dermatitis; atopic dermatitis; contact dermatitis
MeSH Terms: conditions — Dermatitis; Dermatitis, Atopic; Dermatitis, Contact

STUDY DESIGN:
Intervention Model Description: Multicenter, open label, uncontrolled, single arm, post-market clinical folow-up study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DermoRelizema ecofoam (Experimental): DermoReizema ecofoam for 42 days, 2 times per day
  Interventions: Device: DermoRelizema ecofoam

INTERVENTIONS:
Device: DermoRelizema ecofoam — DermoRelizema ecofoam, class II a medical device, topical compact mousse, to be applied 2 times per day during the 42 days of study duration

SUMMARY:
The scope of this open label clinical trial is to evaluate and confirm the performance of DermoRelizema ecofoam in the improvement of the dermatitis severity, by alleviating the symptomatology. The disease severity will be clinically measured through the Investigator Global Assessment (IGA) after 28 days of treatment.

DETAILED DESCRIPTION:
The scope of this open label clinical trial is to evaluate and confirm the performance of DermoRelizema ecofoam in the improvement of the dermatitis severity, by alleviating the symptomatology. The product will be applied for 42 days of treatment, 2 times per day into the face.

The dermatologist will perform 3 clinical follow up visits to assess the efficacy and safety of the product

ELIGIBILITY:
Inclusion Criteria:

1. Subject's written informed consent obtained prior to any studyrelated procedures;
2. Generally healthy male and female aged ≥ 18 years;
3. Presence of dermatitis of any typology, including atopic dermatitis (AD), irritant contact dermatitis (ICD) or allergic contact dermatitis (ACD), of mild-moderate severity:

   * IGA score 2 (=mild) or 3 (=moderate);
4. Dermatitis affecting one or more body areas (face, legs, arms, etc.);
5. Subjects with cooperative attitude, able to comprehend the full nature and the purpose of the investigation, including possible risks and side effects, and able to comply with the requirements of the entire investigation (including ability to attend the planned visits according to the time limits), based on Investigator's judgement.

Exclusion Criteria:

1. Severe dermatitis at inclusion;
2. Pregnant and breastfeeding women;
3. Concomitant other skin disorders including skin infections;
4. Currently or previously diagnosed or treated (chemotherapy and/or radiotherapy) for cancer in the past 5 years;
5. History of previous skin cancer (history of non-metastatic squamous or basal cell carcinoma of the skin is allowed);
6. Active infections or use of antibiotics in the past 7 days;
7. Diabetic subjects;
8. History of congenital or acquired immunodepression;
9. Immunologic or infectious disease (e.g. hepatitis, tuberculosis, HIV or AIDS, any typology of lupus, rheumatoid arthritis) which could place the subject at risk or interfere with study results;
10. Use of any topic medication for dermatitis in the past 14 days;
11. Use of any topic product for dermatitis in the 2 days before study treatment start;
12. Any systemic treatment or procedure that could influence dermatitis activity within the past 30 days (or 5 half-lives);
13. Use of any corticosteroids, immunosuppressant drugs or immunotherapy within the past 30 days (or 5 half-lives);
14. Use of oral antihistamines and antidepressants in the past 30 days;
15. Subjects with any other clinically significant or unstable concurrent disease or skin condition or general condition that, in the Investigator's opinion, might interfere with the study evaluations;
16. Allergy, sensitivity or intolerance to the components of the investigational device formulations ingredients;
17. Concomitant or previous participation in other interventional clinical study in the past 3 months;
18. Subjects planning sun exposure or tanning booths or UV sources throughout the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Fabbrocini, MD, Principal Investigator — Ospedale "Federico II" Napoli
Locations (1):
- Azienda Ospedaliero Universitaria "Federico II", Napoli, Italia, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 40 subject were enrolled in the study, signed the informed consent forms, attended the first visit and 40 started the treatment. Among them, 6 subjects withdrew from the study between V1 and V4 ( 3 subjects because they needed to start a not allowed medication, 2 were lost to follow-up and 1 withdrew the consent). Based on this, 34 subjects, out of 40, regularly completed the study.
Period: Overall Study
Arm/Group | DermoRelizema Ecofoam
Started | 40
Completed | 34
Not Completed | 6
Not completed — Lost to Follow-up | 2
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The demographic characteristics were analysed on FAS population
Groups:
- DermoReizema Ecofoam for 42 Days, 2 Times Per Day: DermoRelizema ecofoam is a topical compact mousse, to be applied 2 times per day, the first application in the morning and the second in the evening before bed time, for 42 consecutive days.
Arm/Group | DermoReizema Ecofoam for 42 Days, 2 Times Per Day
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 37
Region of Enrollment [Number; unit: participants]
  Italy | 37
Number of partecipants with clinical diagnosis of dermatitis of mild-moderate severity:IGA score 2-3 [Number; unit: participants] — IGA (Investigator Global Assessment) is a six-point scale (0 = clear, 1 = almost clear, 2 = mild, 3= moderate, 4 = severe, 5 = very severe.
  participants | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Partecipants With Improvement of Dermatitis Severity
Description: The primary endpoint was the change from baseline ( visit 1) to day 28 ( visit 3) in Investigator Global Assessment (IGA) and the assestment was also dichotomized in terms of treatment success or treatment failure
Time Frame: 28 days of treatment
Population: Primary endpoint data was analyzed in the FAS population and the analysis was then repeated in the PPAS population
Measure: Count of Participants; unit: Participants
Arm/Group | DermoRelizema Ecofoam
Number analyzed (Participants) | 37
Participants | 37

2. Secondary Outcome: Percentage of Partecipants With Improvement of the Dermatitis Severity
Description: to evaluate the performance of the DermoRelizema ecofoam in the improvement of dermatitis severity (IGA) after 14 and 42 days of treatment;
Time Frame: after 14 and 42 days of treatment
Population: This endpoint was conducted on the FAS population
Measure: Count of Participants; unit: Participants
Arm/Group | DermoRelizema Ecofoam
Number analyzed (Participants) | 37
Participants | 35

3. Secondary Outcome: Eczema Area and Severity Index Scores
Description: to evaluate the eczema improvement through the EASI (Eczema Area and Severity Index) score. Severity strata for the EASI were as follows: 0 = clear; 01-1.0 = almost clear; 1.1-7.0 = mild; 7.1-21.0 = moderate; 21.1-50.0 = severe; 50.1-72.0 = very severe
Time Frame: to 14, 28 and 42 days of treatment
Population: EASI score change from baseline to every following time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DermoRelizema Ecofoam
Number analyzed (Participants) | 37
units on a scale
  baseline | 2.60 (1.94)
  after 14 days | 1.20 (1.03)
  after 28 days | 0.80 (1.32)
  after 42 days | 0.20 (1.33)

4. Secondary Outcome: VAS Scores for Itcing, Burning, Pain and Prurits at Visits
Description: to evaluate the improvement in pain and pruritus at visits, as reported by the subject at visits by VAS (Visual Analogue Scale). The subject was requested to indicate at each visit his/her pruritus, itching, burning and pain by placing a vertical mark along a 100 mm VAS (Visual Analogue Scale). The rating was recorded as a distance from the left side of the scale (0 mm) to the mark made by the patient.
Time Frame: to 14, 28 and 42 days of treatment
Population: Change in ichting, burning, pain and prurits by VA from baseline to every following time point was analized using paired student's t-test if the variable is normally distribuited and wilcoxon signed rank test if the variabile is not normally distribuited. The subject was requested to indicate at each visit his/her pruritus, itching, burning and pain by placing a vertical mark along a 100 mm VAS (Visual Analogue Scale). .
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | DermoRelizema Ecofoam
Number analyzed (Participants) | 37
score on a scale
  itching at baseline | 32.00 (30.09)
  itching at day 14 | 17.00 (23.29)
  itching at day 28 | 3.00 (12.33)
  itching at day 42 | 16.46 (0.00)
  burning at baseline | 24.00 (27.24)
  burning at day 14 | 18.40 (10.50)
  burning at day 28 | 8.69 (2.00)
  burning at day 42 | 0.00 (11.95)
  pain at baseline | 4.00 (20.29)
  pain at day 14 | 0.00 (12.58)
  pain at day 28 | 0.00 (12.17)
  pain at day 42 | 0.00 (4.43)
  pruritus at baseline | 52.00 (31.60)
  pruritus at day 14 | 24.00 (26.98)
  pruritus at day 28 | 10.00 (15.24)
  pruritus at day 42 | 1.00 (19.38)

5. Secondary Outcome: Percentage of Partecipants With Improvement in the Quality of Life (QoL)
Description: to evaluate improvement in the Quality of Life (QoL) of the subject related to his/her dermatitis, through the DLQI (Dermatology Life Quality Index) questionnaire; DLQI is a questionnaire used to measure the impact of skin disease on the quality of life of an affected person. There are 10 questions, covering the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, treatment. Each question refers to the impact of the skin disease on the patient's life over the previous week.
  Each question was scored from 0 to 3, giving a possible score range from 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life).
  Global score:
  0-1 = No effect on patient's life 2-5 = Small effect 6-10 = Moderate effect 11-20 = Very large effect 21-30 = Extremely large effect.
Time Frame: to 14, 28 and 42 days of treatment
Reporting Status: Not Posted

6. Secondary Outcome: Number of Partecipants With Adherence to Treatment.
Description: number of partecipants with adherence to treatment.
Time Frame: to 14, 28 and 42 days of treatment
Population: The subject's adherence to treatment was assessed through the number of applications reported on the subject's diary.
Measure: Number; unit: number of partecipant
Arm/Group | DermoReizema Ecofoam for 42 Days, 2 Times Per Day
Number analyzed (Participants) | 37
number of partecipant | 36

7. Secondary Outcome: Percentage of Patient With Improvement of Performance by IGA
Description: to evaluate the subject's and Investigator's global evaluation of performance of DermoRelizema ecofoam by means of a 7-items scale (where 1 = very much improved, 2 = improved, 3 = minimally improved, 4
  = no change, 5 = minimally worse, 6 = worse, 7 = very much worse)
Time Frame: at the end of the study ( day 42)
Measure: Count of Participants; unit: Participants
Arm/Group | DermoReizema Ecofoam for 42 Days, 2 Times Per Day
Number analyzed (Participants) | 37
Participants | 36

8. Secondary Outcome: Percentage of Partecipants Who Indicated That the Treatment Was Acceptable
Description: to evaluate the subject's overall acceptability of the treatment (which takes into account pleasant or unpleasant feeling with the product and the ease of use), performed by means of a 5-item scale (where 1 = very much satisfied, 2 = satisfied, 3 = neither satisfied nor dissatisfied, 4 = dissatisfied, 5 = very much dissatisfied)
Time Frame: at the end of the study ( day 42)
Population: the acceptability was obteined by means of a 5 item scale will be summarized through number and the proportion of subject for each item
Measure: Number; unit: percentage of participants
Arm/Group | DermoReizema Ecofoam for 42 Days, 2 Times Per Day
Number analyzed (Participants) | 37
percentage of participants | 83.8

ADVERSE EVENTS:
Time Frame: All subject enrolled were treated with DermoRelizema ecofoam for 42 consecutive days
Description: Only two adverse event were registred during the study. This events were not related to the study treatment
Arm/Group | DermoRelizema Ecofoam
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 2/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DermoRelizema Ecofoam (N=40)
Infection (Infections and infestations) | 1 — COVID 19 infection
erythema with vesiculation and pruritus (Skin and subcutaneous tissue disorders) | 1 — Worsening of clinical manifestations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/71/NCT04826471/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT04826471/SAP_001.pdf